CLINICAL TRIAL: NCT00410878
Title: A Repeated-Dose Pharmacokinetic Evaluation of Dilaudid SR Tablets (Hydromorphone HCI) in Patients With Chronic Pain
Brief Title: A Repeated Dose Study of the Metabolism and Action Evaluation of OROS Hydromorphone HCI (Slow Release) Tablets in Patients With Chronic Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alza Corporation, DE, USA (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR011620
Record Dates: First submitted 2006-12-12; First posted 2006-12-13 (Estimated); Last update posted 2017-02-17 (Actual); Status verified 2010-04

CONDITIONS: Pain; Analgesics, Opioid
Keywords: Opioids; Chronic cancer pain; Analgesic
MeSH Terms: conditions — Pain

INTERVENTIONS:
Drug: OROS Hydromorphone HCI (slow release)

SUMMARY:
The purpose of this study was to characterize the steady-state pharmacokinetic (metabolism and action) profile of OROS hydromorphone HCI (slow release) in patients who required opioid therapy on a daily basis for chronic pain conditions. Patients stabilized on prior opioids were converted to OROS hydromorphone slow release and titrated (slowly increased or decreased) to adequate analgesia (pain relief). They were maintained at that dose for 4-10 days and had blood samples drawn over 24 hours on the last day of study.

DETAILED DESCRIPTION:
This was an open-label, repeated-dose study involving patients who required opioid therapy on a daily basis for chronic pain conditions. In this study, baseline evaluations were performed at Visit 1. Patients were given a diary in which to record daily opioid medication use and daily pain-relief ratings throughout the study. During the time between Visit 1 and Visit 2 patients continued taking their prior oral or transdermal opioid medication for pain. Patients were considered stabilized when during usual activity, the total daily dose of baseline medication remained unchanged, with no more than three opioid breakthrough pain medication doses/day administered, for two consecutive days. Patients returned within 1 week of Visit 1 for Visit 2. During this visit, patient's 24-hour baseline oral opioid dose was converted to hydromorphone at a conversion ratio of approximately 5:1 (oral morphine sulfate to oral hydromorphone HCI mg equivalents). Patients were dispensed OROS hydromorphone HCI slow release tablets and were then increased to acceptable analgesia (pain relief). Eligible stabilized patients requiring a total daily dose of at least 8 mg but no more than 64 mg of OROS hydromorphone HCI slow release (exclusive of breakthrough medication) began the 5-10 day maintenance therapy phase at Visit 3. Morphine sulfate (immediate-release tablets) were provided as breakthrough pain medication. Patients returned to the clinic in the morning following a minimum of 4 days of continuous OROS hydromorphone HCI slow release therapy at a constant daily dose for Visit 4. Upon arrival at the clinic, an initial (trough) blood sample was taken prior to witnessed administration of the usual dosage of OROS hydromorphone HCI slow release. The exact time of the drug administration was documented. Patients were instructed to return the following morning and not to consume food or beverage within 3 hours of their scheduled visit. Patients were instructed not to self administer their OROS hydromorphone HCI slow release the following morning; they were dosed in the clinic. Patients could take immediate release morphine sulfate as needed. Patients returned to the clinic the next morning (visit 5) and remained for a 24-hour period for witnessed dosing and plasma (blood) sampling for pharmacokinetic (metabolism/action) analysis. Dosing and plasma (blood) sampling began 24 hours following the time of dosing at the clinic the previous day. Water (240 mL) was taken with the medication. Immediately prior to each blood draw, patients rated their pain intensity using an 11-point scale and rated their pain intensity from 0 (no pain) to 10 (pain as bad as you can imagine). Blood samples for analysis were drawn at: 0 (prior to dosing), 1,2,4,6,8,10,12,15,18,21 and 24 hours after dosing. Urine output was collected over the 24-hour period from selected patients. Vital signs were taken. At the conclusion of Visit 5 or in the event of early study termination, a Global Evaluation and physical examination were performed. The patient's diary was reviewed with the patient and all unused study medication was collected. Safety assessments included vital signs and physical examination at the start and end of study. OROS Hydromorphone HCL (slow release) 8,16,32,and 64 mg tablets orally. Patients were stabilized on prior opioids then converted to OROS Hydromorphone HCL (slow release) and slowly increased or decreased to adequate analgesia. Then the patients were maintained at that dose for 4 - 10 days. Duration of treatment was up to 31 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had chronic nonmalignant or chronic cancer pain and were currently receiving strong oral or transdermal opioid analgesics (drug that relieves pain) on a daily basis or patients suitable for advancement of therapy to step 3 on the WHO (World Health Organization) analgesic (drug that relieves pain) ladder
* Patients who required the opioid equivalent of at least 32 mg but no more than 300 mg of oral morphine sulfate or opioid equivalent (exclusive of breakthrough pain medication) every 24 hours for the management of chronic nonmalignant or cancer pain
* Patients who were expected to have reasonably stable opioid requirements for the duration of the study

Exclusion Criteria:

* Patients intolerant of or hypersensitive to hydromorphone (or other opioid drugs)
* Patients who were pregnant or breast-feeding.Patients with any dysphagia or unable to swallow tablets, acute abdominal conditions that may be obscured by opioids or gastrointestinal disorders, including pre-existing severe GI narrowing, that may affect the absorption or transit of orally administered drugs
* Patients with any significant CNS disorder, including but not limited to head injury, intracranial lesion, increased intracranial pressure, seizure disorder, stroke within the past 6 months, and disorders of cognition, and clinically significant impaired hematological function
* Patients that may be at risk for serious decreases in blood pressure following administration of an opioid analgesic (pain relief)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Study Completion 1999-08 (Actual)

PRIMARY OUTCOMES:
The pharmacokinetic (absorption, distribution, excretion) profile of OROS hydromorphone. The time required for absorption and distribution in the body.

SECONDARY OUTCOMES:
Relationships between pharmacokinetic (absorption, distribution, excretion) and pharmacodynamic (drug action on body systems) responses. Patients rated their pain intensity prior to each time blood was draw.

CONTACTS AND LOCATIONS:
Overall Officials: Alza Corporation Clinical Trial, Study Director — ALZA